CLINICAL TRIAL: NCT05780853
Title: Evaluation of a Novel Game-based Neurodevelopmental Assessment for Young Children
Brief Title: A Game-based Neurodevelopmental Assessment for Young Children
Acronym: BRIGHTEN
Status: Recruiting | Type: Observational
Sponsor: Brightlobe Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: BRIGHTEN-01
Record Dates: First submitted 2023-02-10; First posted 2023-03-23 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Neurodevelopmental Disorders; Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder; Dyslexia; Specific Learning Disorder; Child Development
Keywords: Diagnostic test; Neurodevelopment; Medical technology
MeSH Terms: conditions — Neurodevelopmental Disorders; Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Dyslexia; Specific Learning Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Typically Developing Children (Control Group): Typically developing children with no known neurodevelopmental disorder, medical comorbidities, a chronic illness or any additional diagnoses that would impact their ability to complete the game-based assessment.
  Interventions: Diagnostic Test: Tablet Game-based Assessment - YARN assessment service; Diagnostic Test: Adaptive Behavior Assessment System, Third Edition (ABAS-3); Other: Demographic questionnaire
- Children with a Diagnosed Neurodevelopmental Disorder (Clinical Group): Children with a diagnosed neurodevelopmental disorder including: Attention Deficit Hyperactivity Disorder (ADHD), Autism Spectrum Disorder (ASD), Specific Learning Disorder, or a Communication Disorder. Children must also have no known medical comorbidities, a chronic illness or any additional diagnoses that would impact their ability to complete the game-based assessment.
  Interventions: Diagnostic Test: Tablet Game-based Assessment - YARN assessment service; Diagnostic Test: Adaptive Behavior Assessment System, Third Edition (ABAS-3); Other: Demographic questionnaire

INTERVENTIONS:
Diagnostic Test: Tablet Game-based Assessment - YARN assessment service — Tablet game-based assessment to assess neurodevelopmental profile.
Diagnostic Test: Adaptive Behavior Assessment System, Third Edition (ABAS-3) — A parent-reported child behavioural assessment questionnaire used to diagnose and classify various developmental, learning and behavioural disabilities and disorders.
Other: Demographic questionnaire — Parent/carer and child's demographic data such as age, ethnicity, employment status, household income, medical history and education status.

SUMMARY:
The aim of this study is to evaluate a novel tablet game-based neurodevelopmental assessment tool for young children aged 3 to 8 years old.

The study's main aims are: (1) to determine whether the novel tablet-game based assessment tool can accurately differentiate children's neurodevelopmental status based on their performance on the game and (2) assess the validity of the game-based neurodevelopment assessment tool.

The study aims to recruit 590 children who are 'typically' developing and/or have a diagnosed neurodevelopmental disorder including Attention Deficit Hyperactivity Disorder (ADHD), Autism Spectrum Disorder (ASD), Specific Learning Disorder, or a Communication Disorder.

All participants will complete the tablet game-based assessment which aims to assess a range of neuropsychological functions including attention, memory, language, motor, executive functions and social-emotional skills. Parents/carers of participants will also complete a demographic questionnaire and the Adaptive Behaviour System - Third Edition (ABAS-3), which is a questionnaire that assesses a child's development. Some participants will be re-tested on the tablet game-based assessment approximately 2 weeks after the first tablet game-based assessment to ensure the game's validity.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 8 year old 'typically' developing children with no known neurodevelopmental disorder.

OR

* 3 to 8 year old children with a diagnosed neurodevelopmental disorder, including Attention Deficit Hyperactivity Disorder (ADHD), Autism Spectrum Disorder (ASD), Specific Learning Disorder, or a Communication Disorder.

All parents/caregivers and children must have a minimum level of English fluency required to complete the parent questionnaire and the game-based assessment.

Exclusion Criteria:

* Children with medical comorbidities, a chronic illness or any additional diagnoses that would impact their ability to complete the game-based assessment.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children will be recruited into the study from nurseries, preschools, infant and primary schools across the United Kingdom. The study will also be shared across local libraries, playgroups, online parenting forums and groups, and parent-specific publications to make parents aware of the study.
Sampling Method: Non-Probability Sample
Enrollment: 590 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the tablet game-based assessment | 16 months
  Sensitivity and specificity of the tablet game-based assessment to accurately differentiate children's neurodevelopmental status.
Construct validity of the tablet game-based assessment | 16 months
  Using exploratory factor analysis to explore the construct validity of the tablet game-based assessment.
Internal consistency of the tablet game-based assessment | 16 months
  Cronbach's alpha and omega statistic to assess internal consistency/reliability of the tool, which assesses the extent to which all the items in the game-based assessment measure the same concept or construct.
Known-group and predictive validity of the tablet game-based assessment | 16 months
  Known-group and predictive validity will both be assessed through multiple logistic regression.

SECONDARY OUTCOMES:
Preliminary normative data for performance on the tablet game-based assessment tool | 16 months
  Performance on the tablet game-based assessment tool will be obtained from metadata and psychometric data obtained from the game-based assessment tool and device such as response time, correct/incorrect responses and gyroscope readings. Performance scores may be dichotomous, continuous and/or counts. Preliminary normative data for performance on the tablet game-based assessment tool will be defined through an exploratory factor analysis.
Acceptability of the tablet game-based assessment tool and device | 16 months
  Parent and child acceptability of the tablet-game based assessment tool and device will be conducted by asking parents 3 brief questions to assess parental perception of acceptability (e.g. Having seen your child complete the game today, how do you think they found the experience?). Child acceptability will be accessed using a smileyometer scale (5 ratings) to rate how they felt about the game-based assessment. Children will also be asked 8 brief questions about their opinions on the game (e.g. What did you think about the game?).
Re-test reliability of the tablet game-based assessment tool | 16 months
  Acceptable levels of test-retest reliability/stability using Intraclass Correlation Coefficient (ICC) at two different time points within 2 weeks.
Safety of the tablet game-based assessment tool and device | 16 months
  Any adverse events occurring during the duration of the study will be recorded and reported at the end of the study. These will be recorded as the number of events with qualitative data about the nature of the event. These events will then be grouped into different types of risk, and how likely they would be to occur in any future use of the device.

OTHER OUTCOMES:
Participant demographics | 16 months
  Descriptive analyses of participant demographics (e.g., age, ethnicity, employment status, household income, medical history and education status)
Scores on the Adaptive Behavior Assessment System, Third Edition (ABAS-3) | 16 months
  Scores on the parent-reported questionnaire (ABAS-3)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Iles, PhD DClinPsy, Principal Investigator — Brightlobe Limited
Locations (1):
- Brightlobe Limited, London, United Kingdom